CLINICAL TRIAL: NCT01410526
Title: Assessment of Peritoneal Immune Response in Patients With Severe Intra-abdominal Sepsis Managed With Laparostomy and Vacuum Assisted Closure (VAC)
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Associate Professor in Surgery, Aristotle University Of Thessaloniki
Other Study IDs: 1354_9/5/2011
Record Dates: First submitted 2011-07-05; First posted 2011-08-05 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Abdominal Sepsis
Keywords: VAC; Severe abdominal sepsis; Peritoneal immune reaction; Peritonitis; Immune peritoneal reaction when abdominal sepsis is treated with VAC
MeSH Terms: conditions — Intraabdominal Infections; Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- VAC group: Patients with intra-abdominal sepsis treated with Vacuum Assisted Closure (VAC) system plus the dynamic sutures
- Control group: Patients suffering major abdominal surgery

SUMMARY:
Protocol Synopsis

Protocol title: Assessment of peritoneal immune response in patients with severe intra-abdominal sepsis managed by laparostomy and VAC

Purpose: Assessment of peritoneal immune response in patients with severe intra-abdominal sepsis

Design: Prospective, single-center study

Patient Population: Male or female adults (>18 years) with severe intra-abdominal sepsis

No. of Subjects: 60 patients divided into two groups, 30 patients with severe intra-operative sepsis and 30 patients without sepsis scheduled to undergo major abdominal operations (middle line incision>15cm). The study is estimated up to 2 year to enroll

Duration of Follow-up: Follow-up will be performed daily while hospitalized, until patient discharged or deceased.

Endpoints:

1. To measure the peritoneal cytokines levels in patients with severe intra-abdominal sepsis.
2. To correlate the cytokines levels in the abdominal cavity and the serum plasma.
3. To correlate cytokines response in serum plasma and peritoneal fluid with mortality and morbidity.
4. To compare cytokines results in serum plasma and peritoneal fluid between patients with severe intra-abdominal sepsis and patients undergoing major laparotomy without sepsis.
5. To assess the microbial load in the abdominal cavity in patients with severe sepsis.
6. To assess the biofilm formation in VAC polyurethane sponge.

DETAILED DESCRIPTION:
Principal Investigator Statement: ……………………………………………… 1 Protocol Synopsis: ……………………………………………………………… 2 Table of Content: ………………………………………………………………. .4 1.0 Introduction: ……………………………………………………………. 5 2.0 Techniques descriptions: ……………………………..………………… 6 3.0 Objectives: ……………………………..…………………………………7 4.0 Design and study population: …………………………………………… 7 5.0 Study procedure: ……………………………..………………………… 8 6.0 Complications and adverse events: …………………………………… 15 7.0 Statistical analysis: ……………………………..……………………… 15 8.0 Data monitoring plan: ……………………………..………………… 16 9.0 Data confidentiality: ……………………………..…………………… 16 10.0 Funding: ……………………………..………………………………… 16 11.0 Ethics: ……………………………..…………………………………… 16 12.0 Informed consent: ……….……………………………..………………. 17 13.0 References: ……………………………………..……………………… 18

1.0 INTRODUCTION

Severe abdominal sepsis is defined as sepsis plus organ dysfunction caused by a condition deriving from the peritoneal cavity [1]. The essentials of the management of patients with severe sepsis remain unchanged and can be divided broadly into sepsis control, antimicrobial therapy and hemodynamic stabilization [2]. Infection control mainly involves surgical exploration and temporary or permanent resolution of the septic agent [3]. Open abdomen treatment remains one of the most valid approaches of patients with severe abdominal sepsis [4]. Open abdomen management is mandated to avoid abdominal compartment syndrome, in cases with inability to re-approximate the abdominal fascia regardless to viscera oedema and intra-abdominal pressure and in cases with unclear or inadequate source control [5]. Topical negative pressure with the abdominal vacuum-assisted closure (VAC) device has been introduced, providing a new option to manage an open abdomen [6-8].

Cytokines are a group of proteins produced by a variety of cells playing an active role in the immune system. Sepsis syndrome seems to result from overwhelming systemic inflammation which is caused by excessive release of cytokines into systemic circulation [9]. During the last decade many clinical studies assess the cytokines concentration in serum plasma in patients with SIRS and sepsis [10-13]. Despite the board study and analysis of cytokines response in serum plasma, literature is poor about peritoneum immune response in intra-abdominal sepsis [14-15], whereas the majority of these studies concerned patients with elective surgery [16-18].

This protocol is designed to assess the cytokines levels in the peritoneal cavity in severe intra-abdominal sepsis and to compare these levels with the corresponding values in serum plasma. Additionally, the cytokines values in serum plasma and peritoneum are compared between patients with and without sepsis that underwent major elective laparotomy (middle line incision >15cm). Moreover, cytokines levels are correlated to morbidity and mortality.

2.0 STUDY PROTOCOL In all patients that the origin of sepsis confirmed pre-operative as abdominal, laparotomy will be required. After incision and confirmation of intra-abdominal sepsis, involving the whole peritoneal cavity, peritoneal fluid will be sampled for microbiology culture and cytokines assessment. The appropriate source control interventions will be made and peritoneal lavage will be performed using sterile isotonic sodium chloride solution. At the end of operation a decision for open abdomen will be made by the surgeon, based on the severity of sepsis. If laparostomy will be decided, temporary abdominal closure will be performed with the Vacuum Assisted Closure (VAC) system plus the dynamic sutures [19].

After a two-day application of the VAC, the previous existing dressing will be removed. Peritoneal fluid samples and blood samples will be obtained for cytokines assessment. The abdominal cavity will carefully be rinsed with saline solution and the various abdominal spaces will be inspected for any collections. Additionally, peritoneal fluid sample will be obtained for culture and quantitive analysis. Sequentially, the VAC dressing application will be performed based on previously described protocol [19]. Patients will return to the operating room for sequential fascial closure and replacement of the sponge and sutures every 2 days until the final open abdomen closure. Peritoneal fluid and blood serum samples will be obtained in every VAC change until the permanent abdominal closure or patient's decease. A piece of polyurethane sponge of VAC system will be sent to microbiology department for detection of biofilm formation.

3.0 OBJECTIVES

1. To assess the cytokines in peritoneal fluid in patients with severe intra-abdominal sepsis.
2. To compare the serum plasma cytokines values in patients with severe intra-abdominal sepsis with the corresponding values in the peritoneal fluid.
3. To compare the cytokines values in serum plasma and peritoneal fluid between patients with severe intra-abdominal sepsis and patients without sepsis underwent major elective laparotomy.
4. To evaluate parameters influencing successful, primary abdominal closure, morbidity and mortality.
5. To assess the microbial load in the abdominal cavity in patients with severe sepsis.
6. To assess the biofilm formation in VAC polyurethane sponge.

4.0 DESIGN AND STUDY POPULATION The study is designed as a prospective single center study. Any patient with sepsis suspected pre-operative to be from abdominal origin that will be needed laparotomy and postoperative laparostomy will be assessed.

Control group will be constituted with patients without sepsis that will be underwent major elective laparotomy.

4.1 Inclusion Criteria

1. Patient > 18 years old
2. 30 patients with severe abdominal sepsis in order to form the study group and 30 patients without sepsis undergoing major elective surgery (middle line incision >15cm) to form the control group.
3. Patient or relatives signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

4.2 Exclusion Criteria

1. Patient's Manheim Peritonitis Score < 29
2. Patient's pre-operative SOFA score < 6
3. The use of other temporary abdominal closure system
4. Decease before the first VAC dressing change
5. Patient is participating in another clinical trial which may affect this study's outcomes
6. Patients with immune deficiency
7. Documented seropositivity for human immunodeficiency virus (AIDS)
8. Patient receiving steroids treatment for other medical condition
9. Patient receiving chronic anti-inflammatory treatment
10. Patient receiving anti- TNF treatment
11. Pre-existing parechymal liver disease ( Cirrhosis - Child-Pugh C)
12. Pregnancy

4.3 Duration of the study The study will be conducted until 30 patients of each group are treated. It is estimated that it will take up to 2 year to enroll the patients.

5.0 STUDY GROUP PROCEDURES

5.1 Pre-Surgery

The following pre-surgery information will be recorded:

1. Demographic information including: Date of birth (age), gender, ethnicity
2. Pre-operative duration of sepsis - symptoms
3. Co-morbidities
4. BMI
5. ASA score
6. SOFA score
7. APACHEII score
8. Intra-abdominal pressure (IAP)
9. Preoperative labs (WBC, Ht, Hb, SGOT, SGPT, LDH, Glu, Ure, Cre, K+, Na+, Ca2+, Mg++, TP, Alb, ALP, γ-GT, Amylase)
10. Coagulation (Fibrinogen, PT, aPTT, INR)
11. CRP, PCT, Lectin Binding Protein (LBP)
12. Ischemia Modulated Albumine (IMA)
13. Pre-operative Diagnosis
14. Medications
15. Current and past history of surgical and medical comorbidities
16. Measurement in blood serum plasma sample: IL 1α, IL 1β, IL6, IL8, IL12, IL 10, IL 18, INF-γ, TNF-α, PGF-B, PAF, FGF-β, C5q, C3q, ICAM-I (CD54).
17. Measurement in blood serum plasma sample: fractalkine, CCL6.

5.2 Intra-operative

The surgeon will perform laparotomy and intra-operative sepsis source control. Peritoneal fluid sample will be obtained for culture. Assessment of intra-peritoneal sepsis will be performed and decision for open abdomen management will be made. At the end of the surgery, peritoneal and blood samples will be obtained for cytokines measurement. The following intraoperative variables will be recorded for all patients:

1. Surgery date
2. Operation
3. Manheim Peritonitis Score (MPS)
4. Peritonitis classification (a. fecal peritonitis b. purulent peritonitis, c. necrotizing Pancreatitis, d. postoperative peritonitis, e. necrotizing fasciitis)
5. Procedure relative comments
6. Technical complications
7. Duration of surgery
8. Difficulty of the operation (1=very difficult to 5=very easy)
9. Peritoneal fluid culture
10. Blood serum sample (at closure): (WBC, Ht, Hb, SGOT, SGPT, LDH, Glu, Ure, Cre, K+, Na+, Ca2+, Mg++, TP, Alb, ALP, γ-GT, Amylase, Fibrinogen, PT, aPTT, INR, CRP, PCT, LBP)
11. Blood serum sample (at closure): IL 1α, IL 1β, IL6, IL8, IL12, IL 10, IL 18, INF-γ, TNF-α, PGF-B, PAF, FGF-β, C5q, C3q, ICAM-I (CD54), spectalkine, CCL6.
12. Peritoneal sample (at closure): IL 1α, IL 1β, IL8, IL12, IL 10, IL 18, INF-γ, TNF-α, PGF-B, PAF, FGF-β, C5q, C3q, ICAM-I (CD54), spectalkine, CCL6.

5.3 Admission at Intensive Care Unit (ICU)

1. SOFA Score
2. APACHEII Score
3. Blood serum sample: (WBC, Ht, Hb, SGOT, SGPT, LDH, Glu, Ure, Cre, K+, Na+, Ca2+, Mg++, TP, Alb, ALP, γ-GT, Amylase, Fibrinogen, PT, aPTT, INR, CRP, PCT, LBP)

5.4 Postoperative follow-up

Follow-up evaluation will be performed in every VAC dressing changes while hospitalized in ICU until laparostomy final closure or patient decease. The following information will be recorded for all patients in every change:

1. Assessment of peritoneal cavity
2. Sofa score
3. Peritoneal fluid culture
4. blood serum sample (at change): (WBC, Ht, Hb, SGOT, SGPT, LDH, Glu, Ure, Cre, K+, Na+, Ca2+, Mg++, TP, Alb, ALP, γ-GT, Amylase, Fibrinogen, PT, aPTT, INR, CRP, PCT, LBP)
5. blood serum sample (at change): IL 1α, IL 1β, IL6, IL8, IL12, IL 10, IL 18, INF-γ, TNF-α, PGF-B, PAF, FGF-β, C5q, C3q, ICAM-I (CD54), spectalkine, CCL6.
6. Peritoneal sample (at change): IL 1α, IL 1β, IL6, IL8, IL12, IL 10, IL 18, INF-γ, TNF-α, PGF-B, PAF, FGF-β, C5q, C3q, ICAM-I (CD54), spectalkine, CCL6.
7. Re- operations:
8. Date of re-operation:
9. Re-procedure description :
10. Date of permanent abdominal wall closure:
11. Successful primary abdominal closure: YES NO
12. Type of closure:
13. Duration of open abdomen:
14. Number of VAC dressing changes:
15. Death: YES NO
16. Date of death:
17. Duration of ICU stay:
18. Date of ICU discharge:
19. Duration of hospitalization:
20. Date of discharge:
21. Final patient outcome:
22. Comments

5.5 Blood and peritoneal fluid sampling protocol Blood sample will draw from an indwelling arterial line (10ml) in every VAC dressing change. Aspiration of 5 ml of peritoneal fluid from the Douglas space will be carried out with a syringe prior the lavage. Blood samples allow clotting in glass tubes in room temperature. Peritoneal sample collect in glass tubes. Both blood and peritoneal samples will be centrifuged and the resulting serum will be stored at -70o until processing.

5.6 Bacteriological sampling and cultures At initial explorative laparotomy an aspiration of 5 ml of fluid from the Douglas space will be carried out with a syringe. The sample will be emptied into a rubber membrane-sealed sterile glass tube and will be transported immediately to the laboratory, where it will be directly processed. The same process will be repeated at each change of dressings. Moreover, in every VAC dressing change a piece of the polyurethane sponge will be sent in the microbiology department for detection of biofilm formation.

5.7 Antimicrobic prophylactic regime According to the Greek national guidelines for the antimicrobic therapy, a second generation cephalosporin (750 mg) combined with metronidazole (500 mg) will be empirically used against community acquired peritonitis, 30 minutes prior to induction of anaesthesia. Against postoperative peritonitis, piperacillin-tazobactam (4.5 g) will be employed. The antibiotic schema will be later adjusted according to the peritoneal fluid culture.

5.8 Control group Thirty patients without sepsis scheduled for major elective surgery will constitute the control group. Blood sample and peritoneal fluid sample will be obtained at the end of operation before abdominal closure. Subsequently, blood samples will be obtained at first and third postoperative day for serum plasma cytokines assessment.

Inclusion criteria:

1. Patient is over 18 years old
2. Patient or relatives signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion criteria:

1. Patient is participating in another clinical trial which may affect this study's outcomes
2. Patients with immune deficiency
3. Documented seropositivity for human immunodeficiency virus (AIDS)
4. Patient receiving steroids treatment for other medical condition
5. Pre-existing parechymal liver disease ( Cirrhosis - Child-Pugh C)
6. Pregnancy

6.0 COMPLICATIONS AND ADVERSE EVENTS The coordinator is required to notify the Ethics Committee according to regulations and requirements.

Serious Adverse Events include:

1. Death regardless of cause
2. Any-life-threatening event
3. Any re-hospitalization or prolongation of existing hospitalization
4. Any event that results in persistent or significant disability or incapacity to the patient.

7.0 STATISTICAL ANALYSIS The objective of this study is: a) to assess the peritoneal immune response in patients with severe intra-abdominal sepsis, b) to compare the serum plasma cytokines values in patients with severe intra-abdominal sepsis with the corresponding values in the peritoneal fluid and c) to compare the cytokines values in serum plasma and peritoneal fluid between patients with severe intra-abdominal sepsis and patients without sepsis underwent major elective laparotomy.

Statistical analysis included description of these pre-operative intraoperative and postoperative outcomes, and indication of patient characteristics associated with these outcomes.

In order to efficiently compare the results in patients with severe intra-abdominal sepsis, a control group without sepsis underwent major abdominal surgery was employed (Group A=sepsis and Group B=elective surgery).

Since the study does not have pre-specified hypotheses all statistical analyses are exploratory and interpretation of results should be within this context.

8.0 DATA MONITORING PLAN The coordinator will monitor all data accrual. Furthermore, the coordinator will review the progress of the clinical trial including safety data and ensure as possible that it is conducted, recorded and reported in accordance with the protocol, good clinical practice and the applicable regulatory requirements.

9.0 DATA CONFIDENTIALITY Each patient ill be identified by his/her initials and a unique patient identification number. Source data will be stored with source documents. Only personnel responsible for collecting data and transcribing it into the case report forms will have access to the data. Records will remain on site in secure areas.

10.0 FUNDING No additional funding for the execution of the present protocol is necessary. The investigators are willing to execute the present study without any additional reimbursement.

11.0 ETHICS Prior to study institution review board (IRB) approval should be obtained. Any changes in the study protocol, informed consent forms, or investigator must be re-approved by the IRB. All patients enrolled in the study will provide their consent prior to entering the study. An informed consent form shall be signed and dated by the patient. The investigator will retain the forms as part of the study records.

This study will be executed in accordance with the Declaration of Helsinki, in agreement with the guidelines for conducting a clinical investigation in accordance with the principles of ICH GCP outlined in the E6 document. By signing the present protocol, participants in the study commit themselves to carry it out in accordance with local legal requirements.

12.0 INFORMED CONSENT

All eligible patients or the closest relatives should have the capacity to provide an informed consent.

The above described inclusion and exclusion criteria were designed to ensure the entry of the appropriate population of patients to this study and will be approved by the local IRB. Screening for these criteria will be conducted by the coordinator.

Eligible patients or the closest relatives will be educated about the research proposal by a study investigator. To determine whether the patient or the relatives has understood the issues, he/she will be asked to describe what the research entails and whether they have any questions. All questions will be addressed prior to enrolment. The patient or his legal representative can refuse participation in the study at any time.

A written informed consent form will be generated. For each patient, a case report form (CRF) will be completed, providing general medical information and history.

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years old
2. 30 patients with severe abdominal sepsis in order to form the study group and 30 patients without sepsis undergoing major elective surgery (middle line incision >15cm) to form the control group.
3. Patient or relatives signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures

Exclusion Criteria:

1. Patient's Manheim Peritonitis Score < 29
2. Patient's pre-operative SOFA score < 6
3. The use of other temporary abdominal closure system
4. Decease before the first VAC dressing change
5. Patient is participating in another clinical trial which may affect this study's outcomes
6. Patients with immune deficiency
7. Documented seropositivity for human immunodeficiency virus (AIDS)
8. Patient receiving steroids treatment for other medical condition
9. Patient receiving chronic anti-inflammatory treatment
10. Patient receiving anti- TNF treatment
11. Pre-existing parechymal liver disease ( Cirrhosis - Child-Pugh C)
12. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In all patients that the origin of sepsis confirmed pre-operative as abdominal, laparotomy will be required.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Measure peritoneal immune response to intra-abdominal sepsis | 5/2011-5/2013 (2 years)
  Possible alterations of the following factors in the blood and the periotoneal fluid:
  CRP, PCT, Lectin Binding Protein (LBP),IL 1α, IL 1β, IL6, IL8, IL12, IL 10, IL 18, INF-γ, TNF-α, PGF-B, PAF, FGF-β, C5q, C3q, ICAM-I (CD54),Fractalkine, CCL6.

SECONDARY OUTCOMES:
General characteristics | 5/2011-5/2013 (2 years)
  1. Microbial load in the abdominal cavity.
  2. Biofilm formation in VAC polyurethane sponge.
  3. Characteristics of the patients
  4. Mortality
  5. Morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Michalopoulos, MD, Principal Investigator — 3rd Dpt of Surgery; Theodossis S Papavramidis, PhD, Principal Investigator — 3rd Dpt of Surgery; Spiros Papavramidis, Prof, Study Chair — 3rd Dpt of Surgery; Stella Arampatzi, MD, Principal Investigator — Dpt of Microbiology; Eudoxia Diza-Mataftsi, Prof, Study Chair — Dpt of microbiology; Ioannis Pliakos, MD, Principal Investigator — 3 dpt of Surgery
Locations (1):
- 3rd Department of Surgery, AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] 1.Calandra T, Cohne J. The international sepsis forum consensus conference on definitions of infection in the intensive care unit. Crit Care Med 2005;33:1538-48. 2.Pieracci F, Barie PS. Intrabdominal infections. Curr Opin Crit Care. 2007;13:440-9. 3.Ordoñez CA, Puyana JC. Management of peritonitis in the critically ill patient. Surg Clin North Am 2006;86:1323-49. 4.Stawicki SP, Brooks A, Bilski T et al. The concept of damage control: Extending paradigm to emergency general surgery. Injury 2008;39:93-101. 5.Duff JH, Moffat J. Abdominal sepsis managed by leaving abdomen open. Surgery. 1981;90(4):774-8. 6.Barker DE, Green JM, Maxwell RA, et al. Experience with vacuum-pack temporary abdominal wound closure in 258 trauma and general and vascular surgical patients. J Am Coll Surg 2007;204:784-92 7. Perez D, Wildi S, Demartines N et al. Prospective evaluation of vacuum-assisted closure in abdominal compartment syndrome and severe abdominal sepsis. J Am Coll Surg 2007;205:586-92. 8.Management of the Open Abdomen: From Initial Operation to Definitive Closure. Open abdomen advisory panel: Co-Editors: D. Vargo, J. D. Richardson. Advisory panel: A. Cambell, M. Chang, T. Fabian, M. Franz, M. Kaplan, F. Moore, R. L. Reed, B. Scott, R. Silverman. Am Surg. 2009;75:S1-22. 9.Blackwell TS, Christman JW. Sepsis and cytokines: current status. British J Anaesth. 1996;77:110-7. 10.Oberholzer A, Souza S, Tschoeke S et al. Plasma cytokine measurements augment prognostic scores as indicators of outcome in patients with severe sepsis. Shock. 2005;23(6):488-93.
- [Background] 11.Cogos CA, Drosou E, Bassaris HP et al. Pro-versus anti- inflammatory cytokines profile in patients with severe sepsis: a marker for prognosis and future therapeutic options. J Infect Dis. 2000;181:176-80. 12.Dimopoulou I, Armaganidis A, Douka E et al. Tumour necrosis factor-alpha (TNFa) and interleukin-10 are crucial mediators in post-operative inflammatory response and determine the occurrence of complications after major abdominal surgery. Cytokine 2007;37:55-61. 13.Pettila V, Hynninen M, Takkunen O et al. Predictive value of procalcitonin and interleukin 6 in critically ill patients with suspected sepsis. Intensive Care Med. 2002;28:1220-5. 14.Scheingraber S, Bauerfeilnd F, Bohme J, Dralle H. Limits of peritoneal cytokine measure ements during abdominal lavage treatment for intra-abdominal sepsis. Am J Surg. 2001;18:301-8. 15.Jansson K, Redler B, Truedsson L et al. Intraperitoneal cytokine response after major surgery: higher postoperative intraperitoneal versus systemic cytokine levels suggest the gastrointestinal tract as the major source of the postoperative inflammatory reaction. Am J Surg. 2004;187:372-7 16.Decker D, Tolba R, Spinger W et al. Abdominal surgical interventions: local and systemic conseqouences for the immune system - a prospective study on elective gastrointestinal surgery. J Surg Research. 2005;126:12-8. 17.van Berge Henegouwen M, van der Poll T, van Deventer S, Gouma D. Peritoneal cytokine release after elective gastrointestinal surgery and postoperative complications. Am J Surg. 1998;175:311-6 18.Pedersen M, Qvist N, Bisgaard C et al. Peritoneal microdialysis. Early diagnosis of anastomotic leakage after low anterior resection for rectosigmoid cancer. Scan J Surg. 2009;98:148-54. 19.Pliakos I, Papavramidis TS, Mihalopoulos N et al. Vacuum assisted closure in severe abdominal sepsis with or without retention sutured sequential fascial closure: a clinical trial. Surgery. 2010;148(5):947-53.